CLINICAL TRIAL: NCT00812019
Title: A Phase I/II, Randomized, Observer-blind, Multicenter, Dose Ranging Study to Evaluate the Immunogenicity, Safety and Tolerability of Different Formulations of an Adjuvanted or Non-Adjuvanted Cell Culture-Derived H5N1 Subunit Influenza Virus Vaccine in Healthy Subjects 18 - 40 Years of Age.
Brief Title: Dose Ranging Study to Evaluate Immunogenicity and Safety of Adjuvanted or Non-adjuvanted Cell Culture-derived H5N1 Influenza Vaccine in Young Adults (18-40 Years Old)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seqirus (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V89P1; 2007-003715-32 (EudraCT Number)
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Influenza
Keywords: H5N1 Influenza; Pandemic Flu; MF59 Adjuvant; Cell Culture-Derived; Safety; Immunogenicity; Vaccination; H5N1 influenza pandemic
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- 3.75_0%MF59 (Experimental): Subjects received two 0.5mL vaccinations of cell culture derived H5N1 3.75µg subunit influenza vaccine containing 0% of MF59 three weeks apart.
  Interventions: Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 3.75_0%MF59
- 3.75_25%MF59 (Experimental): Subjects received two 0.5mL vaccinations of cell culture derived H5N1 3.75µg subunit influenza vaccine containing 25% of MF59 three weeks apart.
  Interventions: Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 3.75_25%MF59
- 3.75_50%MF59 (Experimental): Subjects received two 0.5mL vaccinations of cell culture derived H5N1 3.75µg subunit influenza vaccine containing 50% of MF59 three weeks apart.
  Interventions: Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 3.75_50%MF59
- 3.75_100%MF59 (Experimental): Subjects received two 0.5mL vaccinations of cell culture derived H5N1 3.75µg subunit influenza vaccine containing 100% of MF59 three weeks apart.
  Interventions: Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 3.75_100%MF59
- 7.5_0%MF59 (Experimental): Subjects received two 0.5mL vaccinations of cell culture derived H5N1 7.5µg subunit influenza vaccine containing 0% of MF59 three weeks apart.
  Interventions: Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 7.5_0%MF59
- 7.5_25%MF59 (Experimental): Subjects received two 0.5mL vaccinations of cell culture derived H5N1 7.5µg subunit influenza vaccine containing 25% of MF59 three weeks apart.
  Interventions: Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 7.5_25%MF59
- 7.5_50%MF59 (Experimental): Subjects received two 0.5mL vaccinations of cell culture derived H5N1 7.5µg subunit influenza vaccine containing 50% of MF59 three weeks apart.
  Interventions: Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 7.5_50%MF59
- 7.5_100%MF59 (Experimental): Subjects received two 0.5mL vaccinations of cell culture derived H5N1 7.5µg subunit influenza vaccine containing 100% of MF59 three weeks apart.
  Interventions: Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 7.5_100%MF59
- 15_0%MF59 (Experimental): Subjects received two 0.5mL vaccinations of cell culture derived H5N1 15µg subunit influenza vaccine containing 0% of MF59 three weeks apart.
  Interventions: Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 15_0%MF59
- 15_25%MF59 (Experimental): Subjects received two 0.5mL vaccinations of cell culture derived H5N1 15µg subunit influenza vaccine containing 25% of MF59 three weeks apart.
  Interventions: Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 15_25%MF59
- 15_50%MF59 (Experimental): Subjects received two 0.5mL vaccinations of cell culture derived H5N1 15µg subunit influenza vaccine containing 50% of MF59 three weeks apart.
  Interventions: Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 15_50%MF59
- 15_100%MF59 (Experimental): Subjects received two 0.5mL vaccinations of cell culture derived H5N1 15µg subunit influenza vaccine containing 100% of MF59 three weeks apart.
  Interventions: Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 15_100%MF59

INTERVENTIONS:
Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 3.75_0%MF59 — Two vaccinations of Cell Culture-Derived H5N1 3.75 µg Subunit Influenza Vaccine containing 0% of MF59.
  Arms: 3.75_0%MF59
Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 3.75_25%MF59 — Two vaccinations of Cell Culture-Derived H5N1 3.75 µg Subunit Influenza Vaccine containing 25% of MF59.
  Arms: 3.75_25%MF59
Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 3.75_50%MF59 — Two vaccinations of Cell Culture-Derived H5N1 3.75 µg Subunit Influenza Vaccine containing 50% of MF59.
  Arms: 3.75_50%MF59
Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 3.75_100%MF59 — Two vaccinations of Cell Culture-Derived H5N1 3.75 µg Subunit Influenza Vaccine containing 100% of MF59.
  Arms: 3.75_100%MF59
Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 7.5_0%MF59 — Two vaccinations of Cell Culture-Derived H5N1 7.5 µg Subunit Influenza Vaccine containing 0% of MF59.
  Arms: 7.5_0%MF59
Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 7.5_25%MF59 — Two vaccinations of Cell Culture-Derived H5N1 7.5 µg Subunit Influenza Vaccine containing 25% of MF59.
  Arms: 7.5_25%MF59
Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 7.5_50%MF59 — Two vaccinations of Cell Culture-Derived H5N1 7.5 µg Subunit Influenza Vaccine containing 50% of MF59.
  Arms: 7.5_50%MF59
Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 7.5_100%MF59 — Two vaccinations of Cell Culture-Derived H5N1 7.5 µg Subunit Influenza Vaccine containing 100% of MF59.
  Arms: 7.5_100%MF59
Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 15_0%MF59 — Two vaccinations of Cell Culture-Derived H5N1 15 µg Subunit Influenza Vaccine containing 0% of MF59.
  Arms: 15_0%MF59
Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 15_25%MF59 — Two vaccinations of Cell Culture-Derived H5N1 15 µg Subunit Influenza Vaccine containing 25% of MF59.
  Arms: 15_25%MF59
Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 15_50%MF59 — Two vaccinations of Cell Culture-Derived H5N1 15 µg Subunit Influenza Vaccine containing 50% of MF59.
  Arms: 15_50%MF59
Biological: Cell Culture-Derived H5N1 Subunit Influenza Vaccine, 15_100%MF59 — Two vaccinations of Cell Culture-Derived H5N1 15 µg Subunit Influenza Vaccine containing 100% of MF59.
  Arms: 15_100%MF59

SUMMARY:
The aim of the present dose ranging study is to evaluate the safety, tolerability and immunogenicity of two doses of twelve different formulations of a Cell Culture-Derived H5N1 Subunit Influenza Virus Vaccine, adjuvanted with MF59 or non-adjuvanted, given three weeks apart and followed by a booster dose after 12 months in healthy adults 18 to 40 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18-40 years, mentally competent, who have signed an informed consent form after having received a detailed explanation of the study protocol;
* Able to understand and comply with all study procedures and to complete study diaries, to be contacted, and to be available for study visits.

Exclusion Criteria:

* Receipt of another investigational agent within 4 weeks prior to enrollment or before completion of the safety follow-up period in this or in another study; unwilling to refuse participation in another clinical study through the end of this study;
* Receipt of an H5N1 vaccine;
* Receipt of another vaccine within 3 weeks prior to Visit 1 or planned vaccination before Visit 5, or within 3 weeks prior to Visit 7 or before Visit 9;
* Influenza vaccination for the current season within 2 months prior to enrollment (seasonal influenza vaccination is allowed after Visit 5, but no later than 2 months before the booster dose);
* Experience of any acute disease or infection requiring systemic antibiotic or antiviral therapy (chronic antibiotic therapy for urinary tract prophylaxis is acceptable) within 7 days prior to enrollment and prior to the booster dose or fever within 3 days prior to Visit 1 and Visit 7;
* Pregnant or breastfeeding, or females of childbearing potential who refuse to use an acceptable method of birth control during the study period for at least 6 weeks following the booster dose; and, if sexually active, who have not used a reliable birth control method for at least two months prior to study entry;
* Any serious disease, such as: cancer; autoimmune disease; diabetes mellitus type I; diabetes mellitus type II; diabetes relating to genetic defects/syndromes, diseases of the exocrine pancreas or infections; advanced arteriosclerotic disease; moderate or severe chronic obstructive pulmonary disease (COPD); asthma that is greater than mild in severity and/or has exacerbations more than 2 days per week; acute or progressive hepatic disease; acute or progressive renal disease; hyperthyroidism; medically significant bleeding disorders; history of neurological disorders;
* Body mass index (BMI) ≥ 35 kg/m2 where BMI is for obese and not for high muscle mass;
* History of (or current) drug or alcohol abuse, surgery planned during the study period or any other condition that in the investigator's opinion would interfere with safety of the subject or the evaluation of study objectives or the visit schedule;
* Hypersensitivity to any component of the study vaccine;
* Known or suspected impairment/alteration of immune function;
* Members of the research staff or their relatives.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 753 (Actual)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
immunogenicity, safety and reactogenicity of cell culture-derived H5N1 subunit influenza virus vaccines containing different amounts of antigen and adjuvant. | 52 weeks
identification of the optimal adjuvant-antigen dose combination considering antibody titers against the H5N1 strain observed three weeks after two intramuscular doses. | 52 weeks

SECONDARY OUTCOMES:
immunogenicity against heterologous strains of a cell culture-derived H5N1 subunit influenza virus vaccine containing different amounts of antigen and adjuvant. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Scientist, Study Director — Seqirus
Locations (2):
- Baylor College of Medicine, Houston, Texas, United States
- Universitätsklinikum Gießen und Marburg GmbH, Giessen, Germany

REFERENCES:
- [Background] Keitel W, Groth N, Lattanzi M, Praus M, Hilbert AK, Borkowski A, Tsai TF. Dose ranging of adjuvant and antigen in a cell culture H5N1 influenza vaccine: safety and immunogenicity of a phase 1/2 clinical trial. Vaccine. 2010 Jan 8;28(3):840-8. doi: 10.1016/j.vaccine.2009.10.019. Epub 2009 Oct 14. PMID 19835829